CLINICAL TRIAL: NCT05392647
Title: Hetrombopag for Lower-risk MDS With Thrombocytopenia: a Prospective，Open-label, Single-arm Study.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jia Wei, associate chief physician, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-HuB-MDS-II-001
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: hetrombopag; thrombocytopenia; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia | interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Hetrombopag
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — All eligible patients were given hetrombopag orally at an initial dose of 5 mg once daily after overnight fasting (>8 hours of fasting) and at least 2 hours before a meal . The dose of hetrombopag could be modified on the basis of the platelet count of patients after 2 weeks of administration.
  Other Names: Hetrombopag Olamine Tablets

SUMMARY:
The is a phase 2, single-arm, open-label clinical study assessing the efficacy and safety of hetrombopag to increase platelet count in lower-risk MDS patients with thrombocytopenia.

DETAILED DESCRIPTION:
The is a phase 2, single-arm, open-label clinical study assessing the efficacy and safety of hetrombopag to increase platelet count in patients with very low, low, or intermediate risk myelodysplastic syndromes(MDS) according to the revised International Prognostic Scoring System (IPSS-R) with thrombocytopenia. The primary endpoint was proportion of patients achieving platelet response at week 24.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older；
* Confirmed diagnosis of MDS based on 2016 WHO (World Health Organization) and classification with very low, low or intermediate (score ≤ 3.5) risk according to the revised International Prognostic Scoring System (IPSS-R).
* Platelets < 30 x 10^9/L or platelets < 50 x 10^9/L with active bleeding at screening.
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2；
* Ability to understand information material and written informed consent.

Exclusion Criteria:

* Severe active bleeding/infection or any other uncontrolled severe condition;
* History of treatment with thrombopoietin receptor agonists (eltrombopag, avatrombopag, romiplostim, etc.) or recombinant human thrombopoietin with 1 month prior;
* Patients with known active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at screening（If hepatitis B surface antigen or hepatitis B core antibody are positive, HBV-DNA testing are needed. If positive, it suggests a viral replication and subjects will be excluded. If hepatitis C antibody are positive, HCV-RNA testing are needed. If positive, it suggests a viral replication and subjects will be excluded）;
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >2.5 x upper limit of normal (ULN), total bilirubin >2.5 x ULN, creatinine >1.5 x ULN;
* History of portal hypertension or cirrhosis；
* History of any types of solid tumors within 5 years prior, whether the tumors has been treated, metastasized or relapsed (except basal cell carcinoma);
* History of congestive heart failure requiring medical management, cardiac arrhythmias, peripheral arteriovenous thrombosis within 1 years prior, or myocardial infarction or cerebral infarction within 3 months prior;
* ECOG performance score ≥ 3;
* Female subjects who are pregnant or breastfeeding, or subjects who are planning pregnancy within 6 months;
* Women of child-bearing potential and men must agree to use contraception prior to study entry and for the duration of study participation;
* Participated in other clinical trials within 3 months prior;
* Any condition which, in the investigator's opinion, deems the subject an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet response | 24 weeks
  proportion of patients achieving platelet responses at week 24

SECONDARY OUTCOMES:
Overall response rate | 24 weeks
  Patients will be assessed for response according to the IWG criteria.
Proportion of patients with platelet response during treatment | 24 weeks
  Improvement in platelet counts by 24 weeks of therapy
Incidence and severity of bleeding events according to the WHO Bleeding Scale | 28 weeks
  The severity of bleeding symptoms was graded according to the World Health Organization (WHO) bleeding scale (grade 0: no bleeding; grade 1: petechiae; grade 2: mild blood loss; grade 3, gross blood loss; grade 4: debilitating blood loss).
Adverse events | 28 weeks
  Adverse events were recorded and graded according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jia Wei, PhD, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No